CLINICAL TRIAL: NCT07265037
Title: Development of a New Integrated Strategy for Long-Distance and Full-Course Management of Diabetes Using Both Traditional Chinese and Western Medicine: A Combined Online and Offline Approach
Brief Title: Integrated TCM - Western Medicine Strategy for Long - Distance Diabetes Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: YXLL-2025-260
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Integrated Traditional Chinese Medicine and Western Medicine; Telemedicine; Chronic Disease Management; Digital Health
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated TCM-WM Smart Management Group (Other): Participants receive a novel integrated diabetes management strategy via a smart platform (hardware + APP + cloud). This includes TCM-WM baseline assessments, personalized remote monitoring/reminders (glucose, medication, lifestyle), tailored TCM-WM education, and backend multidisciplinary expert support. The management pathway is dynamically optimized every 3 months based on continuous data analysis.
  Interventions: Combination Product: Integrated TCM-Western Medicine Intelligent Diabetes Management Platform
- Conventional Care Group (Other): Participants in this arm receive current standard conventional care for diabetes mellitus. This includes regular outpatient follow-ups by endocrinologists, standard pharmacological therapy (e.g., oral hypoglycemic agents and/or insulin) based on authoritative clinical guidelines such as those from the Chinese Diabetes Society, and routine diabetes health education (e.g., diet and exercise advice) provided by healthcare professionals. Participants in this group do NOT have access to the investigational smart management platform (APP, connected devices), nor do they receive the personalized reminders, remote consultations, integrated TCM-WM management pathway, or proactive management from the backend multidisciplinary team that are part of the intervention. Their care process adheres to the usual practices of their respective medical centers.
  Interventions: Combination Product: Integrated TCM-Western Medicine Intelligent Diabetes Management Platform

INTERVENTIONS:
Combination Product: Integrated TCM-Western Medicine Intelligent Diabetes Management Platform — This intervention is a comprehensive, technology-enabled management strategy. It utilizes an integrated smart platform comprising connected devices (e.g., glucose meters, blood pressure monitors), a mobile application (APP), and cloud services. Participants undergo an initial combined assessment based on Western medicine examinations and Traditional Chinese Medicine (TCM) constitution diagnosis (via questionnaire and tongue image analysis). The platform's algorithms then generate a personalized, automated remote management pathway. This includes customized reminders for monitoring, medication, and follow-ups; tailored lifestyle and health education advice integrating TCM and WM principles; and access to daily online consultations from a backend multidisciplinary expert team (endocrinologists, TCM physicians, nutritionists). The management plan is dynamically optimized every 3 months based on continuous data analysis, forming a closed-loop management system.
  Other Names: Intelligent TCM-WM Diabetes Management System; Digital Integrated Care Platform for Diabetes; Telemedicine-based TCM-WM Collaborative Care; AI-Supported Diabetes Management

SUMMARY:
The management of diabetes is of great value in reducing the risk of complications and alleviating the socioeconomic burden. Currently, the diabetes management models in China have not effectively integrated the advantages of traditional Chinese medicine (TCM) and Western medicine. They also fail to achieve intelligent and automated management, resulting in high management costs and low efficiency. Therefore, it is extremely urgent to explore a new, efficient, convenient, low - cost, and personalized long - distance, full - course, intelligent management model for diabetes that integrates TCM and Western medicine both online and offline.

Based on this, our research group plans to rely on the pre - designed and developed Idata database. We will deeply integrate the diagnostic and treatment advantages of TCM constitution differentiation and Western medical examinations and laboratory tests, construct an automated follow - up path, and build an integrated online diabetes management platform for Internet hospitals, which consists of "intelligent hardware + APP + cloud services + a back - end think - tank of TCM and Western medicine experts + a back - end professional management and care team".

This initiative aims to blaze a new trail in the field of long - distance, full - course, and personalized management of diabetes through the synergy of TCM and Western medicine for Chinese diabetes patients. We expect to significantly reduce the incidence of diabetes complications, remarkably improve the overall health status and quality of life of patients, and bring unprecedented positive impacts on the well - being of diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of typical diabetes symptoms (polyuria, polydipsia, polyphagia, and unexplained weight loss) AND meeting any one of the following laboratory criteria: Fasting venous plasma glucose ≥ 7.0 mmol/L, or Random plasma glucose ≥ 11.1 mmol/L, or Glycated hemoglobin (HbA1c) ≥ 6.5%.
* OR, meeting the following oral glucose tolerance test criteria:Fasting plasma glucose ≥ 7.0 mmol/L AND 2-hour plasma glucose ≥ 11.1 mmol/L after a 75g glucose load.

Exclusion Criteria:

* Comorbidities that may prevent compliance with the study protocol, including but not limited to: active malignancy, rheumatic autoimmune diseases, severe infections, multiple organ failure, or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) | Baseline to 6 Months
  HbA1c reflects average blood glucose levels over the preceding 2-3 months. This outcome measures the absolute change in HbA1c percentage (%) from baseline to the end of the 6-month study period. A larger reduction indicates improved long-term glycemic control.
Percentage of Time in Blood Glucose Target Range (TIR) | Baseline to 6 Months
  Time in Range (TIR) is the percentage of time that a patient's glucose levels remain within a specified target range (3.9-10.0 mmol/L) over a period of time, as measured by continuous glucose monitoring (CGM) or frequent self-monitoring. This outcome assesses the TIR over the entire 6-month intervention period. A higher TIR percentage indicates more stable glucose control and is associated with a reduced risk of diabetes complications.
Glycemic Target Achievement Rate | Baseline to 6 Months
  This outcome measures the proportion of participants who achieve their individualized HbA1c treatment goal (e.g., HbA1c <7.0% for most adults) at the 6-month study endpoint. Achievement is defined based on the latest clinical guidelines and individualized patient factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
The current study protocol does not include a plan to make individual participant data (IPD) publicly available. Data sharing may be considered in the future based on institutional policies and upon reasonable request subject to review and approval.